CLINICAL TRIAL: NCT07232342
Title: Capillary Leak Index Versus Conventional Biomarkers in Predicting Sepsis-Related Outcomes
Status: Recruiting | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, Dr, Benha University
Other Study IDs: BenhaU123456789
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Peritonitis Infectious
Keywords: Peritonitis; Capillary Leak Index; Conventional Biomarkers; Critically Ill Patients
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- adult patients admitted to the ICU with post-operative secondary peritonitis requiring an ICU stay o
  Interventions: Diagnostic Test: Capillary Leak Index Versus

INTERVENTIONS:
Diagnostic Test: Capillary Leak Index Versus — Blood samples will be collected at three time points: within 1-2 hours of ICU admission (Day 0), Day 1, Day 2 and Day 7, to monitor trends in CLI and conventional biomarkers during the ICU stay. • CR

SUMMARY:
This study aims to evaluate the prognostic significance of CLI in predicting 28-day mortality and other outcomes in critically ill patients who develop post-operative abdominal sepsis.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years.

Postoperative secondary peritonitis requiring ICU admission, with clinical evidence of:

Diffuse or localized abdominal pain/tenderness. Peritoneal signs (e.g., guarding, rigidity, rebound tenderness). Imaging or intraoperative confirmation of purulent/exudative intra-abdominal fluid.

Systemic inflammation (e.g., fever, leukocytosis, or vasopressor requirement). Sepsis diagnosis per Sepsis-3 criteria: Suspected/confirmed infection with acute increase in SOFA score ≥2 points (6).

Anticipated ICU stay ≥48 hours postoperatively.

Exclusion Criteria:

* Pregnancy

  * Advanced liver disease (Child-Pugh class B or C) that might independently affect albumin levels
  * Advanced kidney disease (CKD stage 4 or 5) or patients on chronic dialysis
  * Expected mortality within 48 hours of ICU admission
  * Patients with primary peritonitis or tertiary peritonitis
  * Immunocompromised patients (e.g., on chronic immunosuppressive therapy, solid organ transplant recipients, patients with HIV and CD4 count <200/mm³)
  * Patients with pre-existing systemic inflammatory diseases that might affect baseline CRP levels
  * Patients participating in interventional trials that might affect outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients admitted to the ICU with post-operative secondary peritonitis requiring an ICU stay of at least 48 hours will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | From 1-10-2025 to 1-10-2026

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospital, Banhā, Qalyubia Governorate, Egypt